CLINICAL TRIAL: NCT02461862
Title: Assessment of Vital Signs and Pain During Insertion of Intra Uterine Device
Brief Title: Vital Signs and Pain During Insertion of IUD
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Maria Homem de Mello Bianchi, PHD, Federal University of São Paulo
Other Study IDs: Nº CEP: 0272/2015
Record Dates: First submitted 2015-05-25; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Contraception; Acute Pain
Keywords: Contraception; Contraception Behavior; Intra uterine device; Intra uterine System; IUD; IUS; Acute Pain
MeSH Terms: conditions — Acute Pain; Contraception Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Intra Uternine Device: Women who came to the medical service, to insert an intra uterine Device (IUD) of Cu or a Levonorgestrel Intra Uterine System( Lng- IUS) after have been attended in the Family Planning Service of Federal University of São Paulo . All patient have had the pain evaluated by Application of the Visual Analog Scale of Pain (VAS), and also their vital signs ( Evaluation of blood pressure,Evaluation of radial pulse) evaluated pre and five minutes after the IUD/ IUS insertion.
  Interventions: Behavioral: Application of the Visual Analog Scale of pain; Procedure: Evaluation of blood pressure; Procedure: Evaluation of radial pulse

INTERVENTIONS:
Behavioral: Application of the Visual Analog Scale of pain — Evaluation of pain previous and 5 minutes after outpatient insertion of IUD / IUS using the Visual Analog Scale of Pain
  Other Names: VAS
Procedure: Evaluation of blood pressure — Evaluation of Blood pressure ( mmHg), previous and 5 minutes after outpatient insertion of IUD / IUS by sphygmomanometer.
  Other Names: BP evaluation
Procedure: Evaluation of radial pulse — Evaluation of radial pulse (beats per minute) previous and 5 minutes after outpatient insertion of IUD / IUS by pulse oximetry
  Other Names: Pulse evaluation

SUMMARY:
Cross-sectional cohort study to evaluating pain and vital signs variations (blood pressure and radial pulse) during the placement of the intrauterine device.

DETAILED DESCRIPTION:
The intrauterine device (IUD), which is one of the most effective and safe contraceptives is still little used by women. It is considered a long action reversible contraception (LARC). Among the many reasons for this resistance stands the fear of pain, the complications that can occur during the insertion.

Objective: To evaluate the intensity of pain on outpatient insertion of IUD. In addition to evaluating changes in vital signs and detect which are the factors associated with pain on outpatient insertion of IUD. Methods: Cross Sectional Retrospective study of 285 procedures of outpatient insertion of IUD.

Inclusion criteria were age older than 18 years, cervical cytology without abnormalities, classification for Category 1 or 2 of the WHO eligibility criteria for IUD. The criteria for non inclusion were patients with cardiac arrhythmias and gynecological disorders. The insertions of IUD were conducted on an outpatient basis without the use of painkillers.

Evaluation of vital signs ( blood pressure and radial pulse) was performed pre and five minutes after the procedure. The pain assessment was performed using the scale visual analog (VAS), five minutes after the procedure.Correlations of the pain's score with clinical factors as age, parity, BMI, hysterometry, previous vaginal delivery were also performed.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* cytology without abnormalities
* classification for Category 1 or 2 of the WHO eligibility criteria for IUD / IUS.

Exclusion Criteria:

* patients with cardiac arrhythmias
* gynecological disorders

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women that attended to clinical visit to insertion of IUD
Sampling Method: Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain after insertion of IUD/IUS | Single evaluation after 5 minutes of the insertion of the IUD/IUS ( the evaluation takes 1 minute- choose a number on visual analog scale of pain that represents the pain of that moment
  Assessment of pain five minutes immediately after IUD/IUS insertion using the visual analog scale - choose a number on visual analog scale of pain that represents the pain of that moment

SECONDARY OUTCOMES:
Evaluation of blood pressure modification after insertion of IUD/IUS | Duration 15 minutes - two evaluations: before the procedure and five minutes immediately after IUD/IUS insertion
  Evaluation of blood pressure (mmHg) using a Sphygmomanometer, before and five minutes after the insertion of the IUD/IUS
Evaluation of clinical factors that may interfere with the intensity of pain | 1 day
  Correlate the pain score of VAS with clinical factors as age, parity, BMI, hysterometry, previous vaginal delivery
Evaluation of radial pulse modification after insertion of IUD/IUS | Duration 15 minutes - two evaluations: before the procedure and five minutes immediately after IUD/IUS insertion
  Evaluation of radial pulse ( beats per minute) using a pulse oximeter before and five minutes after the insertion of the IUD/IUS

CONTACTS AND LOCATIONS:
Overall Officials: Zsuzsanna IK Jarmy di Bella, Study Chair — Federal University of São Paulo